CLINICAL TRIAL: NCT04834167
Title: OneDoc Picopulse™ for the Treatment of Melasma Among Malaysian Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Yang Mooi Lim, Deputy Director (Institute of Postgraduate Studies and Research), Professor, Universiti Tunku Abdul Rahman
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTAR-45-2021
Record Dates: First submitted 2021-03-24; First posted 2021-04-08 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Skin Diseases; Skin Disorder; Melanoma (Skin)
Keywords: Melasma; Skin treatment; Picopulse; Malaysian women
MeSH Terms: conditions — Skin Diseases; Melanoma; Melanosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Eligible patients will receive ten picopulse treatments for bi-monthly.
  Interventions: Device: OneDoc Picopulse

INTERVENTIONS:
Device: OneDoc Picopulse — Eligible patients will proceed to receive skin cleansing prior to OneDoc Picopulse treatment. After the cleansing, the patients will receive OneDoc Picopulse treatment for 15 mins. Patients will receive ten picopulse treatments for bi-monthly.

SUMMARY:
OneDoc Picopulse™ is a radiopulse technology beauty grade device invented for treating melasma.

DETAILED DESCRIPTION:
This is a new attempt to evaluate the effectiveness of OneDoc PicopulseTM in treating melasma among women of childbearing age in Klang Valley, Malaysia. This pilot feasibility study protocol is to access feasibility of the OneDoc Picopulse™ in the future definitive trial. The findings of this study would justify OneDoc Picopulse™ as one of the promising alternative treatment for melasma.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting dermal melasma with Fritzpatrick skin type III to V
* Malaysian citizen
* Agreed to participate
* Provide informed consent

Exclusion Criteria:

* Patients who had a laser procedure, phototherapy therapy, peel, oral therapy, topical treatment or used lightening creams in the treatment area within the past 6 months.
* Patients with pregnancy, lactating, active dermatitis, had a history of immunosuppression/immune deficiency disorders
* Patients who photosensitivity or taking drugs known to induce photosensitivity,
* Patients that have been exposed to severe sun exposure, having severe epidermal injury, allergy and sensitivity
* Patients who could not attend follow-up treatments

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of the treatment | One month
  Short Assessment of Patient Satisfaction (SAPS) questionnaire with additional Qualitative data collection; The score range for SAPS is from 0 (extremely dissatisfied) to 28 (extremely satisfied)

SECONDARY OUTCOMES:
Feasibility of the recruitment and measurement tools | Pre-treatment, two weeks and one month
  1. Number of patients referred from OneDoc and eligible for screening
  2. Number of patients recruited
  3. Follow-up response rates (2 weeks and 1 month follow-ups)
Treatment adherence | five months
  Number of treatments attended
Melasma | Through study completion, an average of 24 weeks
  Melasma Severity Index (MSI) and by observation; MSI score ranges from 0 (no melasma) to 64 (severe melasma)
Quality of life of patients | Pre-treatment, two weeks and one month post-treatment
  Melasma Quality of Life Scale (MELASQOL) score ranges from 10 to 70; Higher the score, worse is the quality of life
Safety evaluation | immediately after and before each subsequent treatment
  Incidence and severity of side effects caused by treatments

CONTACTS AND LOCATIONS:
Overall Officials: Yang Mooi Lim, PhD, Principal Investigator — Universiti Tunku Abdul Rahman
Locations (1):
- OneDoc, Cheras, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Amini F, Thazin Oo NM, Okechukwu PN, Seghayat MS, Ng ESC. Polymorphisms in P53 and VEGFA genes in different subtypes of periorbital hyperpigmentation in a Malaysian Chinese population. Australas J Dermatol. 2019 May;60(2):e99-e104. doi: 10.1111/ajd.12918. Epub 2018 Sep 14. PMID 30215845
- [Result] Chalermchai T, Rummaneethorn P. Effects of a fractional picosecond 1,064 nm laser for the treatment of dermal and mixed type melasma. J Cosmet Laser Ther. 2018 Jun;20(3):134-139. doi: 10.1080/14764172.2017.1376098. Epub 2017 Dec 4. PMID 29020467
- [Result] Labadie JG, Krunic AL. Long pulsed dye laser with a back-to-back double-pulse technique and compression for the treatment of epidermal pigmented lesions. Lasers Surg Med. 2019 Feb;51(2):136-140. doi: 10.1002/lsm.23009. Epub 2018 Oct 15. PMID 30320904